CLINICAL TRIAL: NCT03313154
Title: Impact on QoL and Cognitive Functioning of New Antiviral Therapies in Subjects With Chronic Hepatitis HCV-related
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria di Cagliari (Other)
Responsible Party: Principal Investigator, Gioia Mura, Dr, Azienda Ospedaliero Universitaria di Cagliari
Other Study IDs: PG/2015/16964
Record Dates: First submitted 2017-09-26; First posted 2017-10-18 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Psychiatric Disorders; Cognitive Impairment; Chronic Hepatitis c
Keywords: Quality of Life; Psychiatric comorbidity; Cognitive impairment; Chronic Hepatitis HCV-related
MeSH Terms: conditions — Mental Disorders; Cognitive Dysfunction; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuropsychiatric screening (treatment+): Subjects affected by chronic hepatitis HCV-related, undergoing new antiviral drugs treatment, will be screened by psychiatric and neuropsychological questionnaires/tests
  Interventions: Other: Neuropsychiatric screening
- Neuropsychiatric screening (treatment-): Subjects affected by chronic hepatitis HCV-related, in wait list for new antiviral drugs treatment, will be screened by psychiatric and neuropsychological questionnaires/tests
  Interventions: Other: Neuropsychiatric screening

INTERVENTIONS:
Other: Neuropsychiatric screening — Psychiatric diagnosis through:
  1. clinical interview
  2. the Advanced Neuropsychiatric Tools and Assessment Schedule (ANTAS), based on the SCID-I-NP (Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders-Non Patient Version);
  3. HAM-D (Hamilton Scale for Depression);
  4. PHQ-9 (Patient's Health Questionnaire-9 items);
  5. MDQ (Mood Disorders Questionnaire);
  6. YMRS (Young Mania Rating Scale);
  7. ASRM (Altman Self Rating Mania scale);
  8. BRIAN (Biological Rhythms Interview of Assessment in Neuropsychiatry).
     Assessment of Quality of Life:
  9. SF-12 (Short Form Health Survey-12 items).
  Neuropsychological screening:
  l) Addenbrooke's Cognitive Examination (ACE-R).

SUMMARY:
Chronic hepatitis HCV-related is the most common cause of chronic liver disease in Italy. Patients with chronic hepatitis C present a prevalence of depressive disorders higher than that of the general population; moreover, it has been repeatedly demonstrated the presence of cognitive deficits and poor quality of life. Chronic hepatitis C therapy was based on the combined use of pegylated alpha-interferons (PEG-INF), and ribavirin. Recently, new therapeutic protocols have been introduced, and while some antiviral drugs, including the first-generation ones, were used only in combination with PEG-IFN and ribavirin, the second and third generation antiviral drugs protocols are interferon-free. However, because of the high cost, the access to interferon-free protocols is only for patients with advanced fibrous stages, or with concomitant extra-hepatic HCV-related diseases, or for transplanted patients. Many side effects, such as flu-like symptoms, and psychiatric symptoms (depression, anxiety, irritability, insomnia) are common during antiviral therapy with IFN. However, in patients with chronic hepatitis C, a high lifetime prevalence of major depressive disorder, panic disorder, and brief recurrent depression have been observed, irrespective of IFN treatment and the use of alcohol and narcotics; such associations between mood and anxiety disorders and chronic hepatitis C may reflect a high prevalence of bipolar spectrum disorders. The presence of severe psychopathological symptoms requires the reduction of posology and causes high rates of discontinuation of antiviral therapy.

This project represents an innovative psychiatric and neuropsychological screening program for patients with chronic hepatitis C, eligible for antiviral therapy.

1. Primary objectives:

   1. to verify the medium-term impact of new antiviral therapies on quality of life, psychological well-being and cognitive function in subjects with chronic hepatitis C;
   2. to verify the predictability of specific psychopathological components and specific determinants on compliance with new antiviral therapies.
2. Main secondary objectives:

   1. to verify the evidence of association between various psychiatric disorders and cognitive deficits and chronic hepatitis C;
   2. to evaluate the relative weight of psychopathological and/or cognitive disorders on the efficacy of antiviral therapy and on quality of life.

DETAILED DESCRIPTION:
Background HCV-related chronic hepatitis represents the most common cause of chronic liver disease in Italy, with an estimated prevalence of 1-1.1% in the general population, reaching about 15% in subjects over 50 years of age. Chronic HCV infection is the cause of 27% of cases of cirrhosis and 25% of cases of hepatocarcinoma. Persons with chronic hepatitis C present a prevalence of depressive disorders higher than that of the general population (59% vs. 21%). Moreover, there has been repeatedly demonstrated the presence of cognitive deficits, mainly concerning attentive, executive, and verbal comprehension, also in the absence of liver cirrhosis and comorbidities due to the use of substances, and a reduced quality of life. Chronic hepatitis C therapy was based on the combined use of pegylated alpha interferons (PEG-INF) and ribavirin, with SVR (sustained virological response, defined as HCV-RNA undetectable in serum at six months after the end of therapy), normalization of transaminases and improvement of liver histology, altogether in 60% of cases. Recently, new antiviral drugs with direct activity (e.g. antiprotease and antipolymer activity) have been introduced into hepatitis C therapeutic protocols, with the development of PEG-INF-free therapeutic schemes. Unfortunately, because of the excessive cost, in many Countries, including Italy, the access to PEG-INF-free schemas is only for patients with advanced fibrous stages, or who have concomitant extra-hepatic viral diseases HCV-related, or those already transplanted, while others are still expected to be treated with PEG-INF and ribavirin.

There are frequent side effects of antiviral therapy, often of minor magnitude, but sometimes incompatible with the continuation of therapy or life threatening. The most common adverse effects are influenza-like symptoms, occurring in more than half of the patients, especially during the first treatment period, and psychiatric symptoms (depression, anxiety, irritability, insomnia), which occur around the third month of treatment from 12 to 41% of patients. However, in persons with chronic hepatitis C, a high lifetime prevalence of major depressive disorder and panic disorder, and brief recurrent depression have been observed, irrespective of PEG-INF treatment and the use of alcohol and narcotic drugs; such associations between mood and anxiety disorders and chronic hepatitis C may reflect a high prevalence of bipolar disorder, which is more difficult to diagnose using non-dedicated screening tools. Some symptoms before treatment start, such as lack of pleasure or interest, asthenia, loss of appetite, social withdrawal, reduced work function, and hostility, are highly predictive of the onset of depressive disorders during antiviral therapy. Poor cognitive performance prior to antiviral therapy, coupled with the only depressive symptom of sadness, is predictive of more severe depressive disorders during antiviral treatment. However, cognitive deficits found before therapy appear potentially reversible and tend to completely recede when there is a virological response sustained by antiviral therapy. The presence of severe psychopathological symptoms leads to a reduction in posology and high rates of discontinuation of antiviral therapy.

Careful psychiatric and neuropsychological evaluation before, during and after antiviral treatment should therefore be an indispensable part of screening and HCV-related chronic hepatitis therapy. This project represents an innovative psychiatric and neuropsychological screening program for persons with chronic hepatitis C, eligible for antiviral therapy. This program aims:

* to determine which psychopathological symptoms and cognitive deficits are more frequent in persons with chronic hepatitis C;
* to verify the impact of antiviral therapy on persons' reported quality of life, and on the onset, aggravation, maintenance of psychopathological symptoms and/or cognitive deficits;
* to determine which psychopathological and neuropsychological symptoms are predictive to high compliance and the effectiveness of antiviral therapy;
* to verify the existence of specific psychopathological and neuropsychological patterns in persons with chronic hepatitis C before, during and after antiviral therapy;
* to produce a standard procedure for psychiatric and neuropsychological screening in patients with HCV-related chronic hepatitis.

Early identification of subjects at risk of psychiatric and cognitive disorders during antiviral therapy will effectively treat individuals at risk of discontinuing the antiviral therapy itself, improving the quality of the treatment and the effectiveness of the treatments.

Design Observational study on a sample of persons with chronic hepatitis C. The experimental cohort will consist of participants who will be admitted to new antiviral treatments. The control cohort will consist of subjects recruited later, for which there is no immediate possibility of access to new treatments (wait-list).

Selection of the sample

The study will be conducted at the Center for the Study of Liver Diseases at the University Hospital of Monserrato, Cagliari. It is intended for subjects with chronic hepatitis C consecutively afferent to the facility, eligible for antiviral therapy. From the whole sample of cases will be drawn two cohorts:

1. approximately 50 subjects with chronic hepatitis C, selected to receive new antiviral therapy immediately;
2. approximately 50 subjects with chronic hepatitis C, who are eligible to receive new antiviral therapy, but are on a waiting list for non-availability of the treatment.

Statistical analysis The data analysis will be carried out after the end of the study and in the next 3 months, by setting up a complete database for each participant, including in an anonymous form the socio-demographic and anamnestic data, and the data from the assessments performed at baseline and in subsequent times. The sample will be analyzed for frequency of lifetime and current psychiatric disorders, current cognitive deficits, subjectively perceived Quality of Life, depressive, hypomanic and manic symptoms, and patterns of biological rhythms. Data analysis will be done with multivariate techniques, for evaluating the effect and interaction of the various factors. The presence of psychiatric disorders and cognitive deficits will be considered dependent variables. The psychopathological specificity of symptoms related to antiviral treatment will also be measured in terms of different frequencies of specific psychiatric/neuropsychological symptoms and specific profiles of response to antiviral therapy. The whole sample will be compared at the baseline with a normative sample extracted with a computerized matching technique (4 controls each case) by gender and age from the database of a Italian population study. Through matchings 1: 4 it will be possible to increase the sample size and increase the statistical power of the study. The data analyses will be performed through SPSS (Statistical Package for Social Science) software.

Funding This project is a spontaneous study, without any source of funding. Ethical Aspects The study will be conducted in accordance with the ethical principles contained in the Helsinki Declaration. The final study protocol was approved by the Ethics Independent Committee of the Azienda Ospedaliero Universitaria di Cagliari (approval record N. PG/2015/16964).

Informed consent The interviewer will give clear and comprehensive information about the nature and the assumptions of the study to the respondents. Participants will also be informed of the possibility of interrupting the interview and withdrawing the consent to the study at any time. Interviewees will be required to sign an informed consent form.

Data protection The subjects enrolled in the study will be given information about data protection and the privacy law. The interviewer will explain that the study data will be placed in a database with anonymous codes to maintain confidentiality, in accordance with local data protection laws.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic hepatitis HCV-related, eligible to new antiviral drugs treatments
* understanding Italian language
* signed informed consent

Exclusion Criteria:

* severe cognitive deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: 50 subjects with chronic hepatitis HCV-related, which are eligible to be immediately treated with new antiviral drugs.
  Group 2: 50 subjects with chronic hepatitis HCV-related, which are eligible to be treated with new antiviral drugs but are in wait list.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Short Form Health Survey-12 item (SF-12) | Baseline (T0), and change from baseline at three (T4) and six (T7) months
  Self-report questionnaire that examines the following dimensions of well-being: vitality, physical function, physical pain, perception of general health, mental, physical, and emotional health, social role.

SECONDARY OUTCOMES:
Advanced Neuropsychiatric Tools and Assessment Schedule (ANTAS) | Baseline (T0)
  semi- structured interview to diagnose most of the psychiatric disorders, consistent with the diagnostic criteria of the DSM IV (Diagnostic and Statistical Manual of Mental Disorders, 4th ed.)
Hamilton Scale for Depression (HAM-D) | Baseline (T0), and change from baseline at three (T4) and six (T7) months
  clinical evaluation scale of the following depressive features: anxiety and somatization, suicidal thoughts, weight loss, cognitive disorders, activity problems, depressive retardation, sleep disturbances, and insight. It consists of 21 items, with scores from 0 to 3. Scoring 8-17 is indicative of mild depression; 18-24 moderate depression; a score> 25 indicates a severe depression.
Patient's Health Questionnaire-9 items (PHQ-9) | Baseline (T0), and change from baseline: at two (T1) and four (T2) weeks, two (T3), three (T4), four (T5), five (T6), and six (T7) months.
  Self-report questionnaire based on the DSM IV Major Depressive Disorder Diagnostic Criteria, investigating the presence and severity in the previous 2 weeks of 9 depressive symptoms, such as depressed mood, anhedonia, sleep and food disorders, fatigue, difficulty concentrating, motor behavior disorders, loss of self-esteem, suicidal ideation; the cut-off for minor depressive disorder is represented by scores ≥5, the one for major depressive disorder by scores ≥10. The questionnaire can be administrated by phone.
Mood Disorders Questionnaire (MDQ) | Baseline (T0)
  Self-report 17-item questionnaire for lifetime screening of bipolar spectrum disorders (Type I and II Bipolar Disorder), through DSM IV diagnostic criteria; the cut-off is for scores ≥7
Young Mania Rating Scale (YMRS) | Baseline (T0), and change from baseline at three (T4) and six (T7) months
  11-item questionnaire, evaluating the severity of manic/hypomanic symptoms (excitement, dysphoria, logorrhea, disorders of form and content of thought, sleep disturbances, aggression, appearance and clothing, insight). A score ≥12 suggests the presence of a manic/hypomanic episode
Altman Self Rating Mania Scale (ASRM) | Baseline (T0), and change from baseline: at two (T1) and four (T2) weeks, two (T3), three (T4), four (T5), five (T6), and six (T7) months.
  self-administered 5-item scale that evaluates the presence and severity in the previous week of manic and hypomanic symptoms, such as manic/irritable mood, increased self-esteem, reduced need for sleep, loquacity, hyperactivity; a score ≥ 6 indicates a high likelihood of a manic or hypomanic episode. It can be administered by phone
Biological Rhythms Interview of Assessment in Neuropsychiatry (BRIAN) | Baseline (T0), and change from baseline at three (T4) and six (T7) months
  21-item questionnaires that investigates the difficulties in sleep, daily activities, social relationships, and nutrition, and how these difficulties relate to biological rhythms
Addenbrooke's Cognitive Examination (ACE-R) | Baseline (T0), and change from baseline at three (T4) and six (T7) months
  short cognitive test, which evaluates five cognitive domains: attention/orientation, memory, verbal fluency, language, visual-spatial abilities. The test, with a maximum score of 100 and a mild cognitive impairment cut-off of 66, includes the Mini Mental State Examination (MMSE).

CONTACTS AND LOCATIONS:
Overall Officials: Gioia Mura, Dr, Principal Investigator — Azienda Ospedaliero Universitaria di Cagliari; Mauro G Carta, Prof, Study Chair — Azienda Ospedaliero Universitaria di Cagliari
Locations (1):
- Policlinico Universitario di Monserrato, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Alter MJ. Epidemiology of hepatitis C virus infection. World J Gastroenterol. 2007 May 7;13(17):2436-41. doi: 10.3748/wjg.v13.i17.2436. PMID 17552026
- [Result] Perz JF, Armstrong GL, Farrington LA, Hutin YJ, Bell BP. The contributions of hepatitis B virus and hepatitis C virus infections to cirrhosis and primary liver cancer worldwide. J Hepatol. 2006 Oct;45(4):529-38. doi: 10.1016/j.jhep.2006.05.013. Epub 2006 Jun 23. PMID 16879891
- [Result] Kraus MR, Schafer A, Faller H, Csef H, Scheurlen M. Psychiatric symptoms in patients with chronic hepatitis C receiving interferon alfa-2b therapy. J Clin Psychiatry. 2003 Jun;64(6):708-14. doi: 10.4088/jcp.v64n0614. PMID 12823087
- [Result] Foster GR, Goldin RD, Thomas HC. Chronic hepatitis C virus infection causes a significant reduction in quality of life in the absence of cirrhosis. Hepatology. 1998 Jan;27(1):209-12. doi: 10.1002/hep.510270132. PMID 9425939
- [Result] Carta MG, Hardoy MC, Garofalo A, Pisano E, Nonnoi V, Intilla G, Serra G, Balestrieri C, Chessa L, Cauli C, Lai ME, Farci P. Association of chronic hepatitis C with major depressive disorders: irrespective of interferon-alpha therapy. Clin Pract Epidemiol Ment Health. 2007 Oct 23;3:22. doi: 10.1186/1745-0179-3-22. PMID 17956625
- [Result] Carta MG, Angst J, Moro MF, Mura G, Hardoy MC, Balestrieri C, Chessa L, Serra G, Lai ME, Farci P. Association of chronic hepatitis C with recurrent brief depression. J Affect Disord. 2012 Dec 10;141(2-3):361-6. doi: 10.1016/j.jad.2012.03.020. Epub 2012 May 18. PMID 22609196
- [Result] Kraus MR, Schafer A, Teuber G, Porst H, Sprinzl K, Wollschlager S, Keicher C, Scheurlen M. Improvement of neurocognitive function in responders to an antiviral therapy for chronic hepatitis C. Hepatology. 2013 Aug;58(2):497-504. doi: 10.1002/hep.26229. Epub 2013 Jun 24. PMID 23300053
- [Derived] Mura G, Chessa L, Manca A, Preti A, Balestrieri C, Onali S, Carta MG. Impact of direct-acting antiviral drugs for chronic hepatitis C on mood: Preliminary results from a longitudinal study. Gen Hosp Psychiatry. 2019 Jan-Feb;56:50-51. doi: 10.1016/j.genhosppsych.2018.10.008. Epub 2018 Nov 14. No abstract available. PMID 30470569